CLINICAL TRIAL: NCT02303184
Title: TANZANITE: Safety and Efficacy of Suprachoroidal CLS-TA in Combination With Intravitreal Aflibercept in Subjects With Macular Edema Following Retinal Vein Occlusion
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide With IVT Aflibercept in Subjects With Macular Edema Following RVO
Acronym: TANZANITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLS1003-201
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: RVO; ME; Central Subfield Thickness; OCT; optical coherence tomography; cystoid macular edema; subretinal fluid; Eylea; aflibercept; anti-VEGF
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — salicylhydroxamic acid; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 mg CLS-TA + IVT aflibercept (Experimental): Single unilateral, suprachoroidal injection of 40 mg/mL (4 mg in 100 µL) of CLS-TA following a 2 mg intravitreal injection of aflibercept
  Interventions: Drug: 4 mg CLS-TA; Drug: IVT aflibercept
- sham + IVT aflibercept (Active Comparator): Single unilateral, suprachoroidal sham procedure following a 2 mg intravitreal injection of aflibercept
  Interventions: Drug: Sham; Drug: IVT aflibercept

INTERVENTIONS:
Drug: 4 mg CLS-TA — 40 mg/mL CLS-TA, Clearside's formulation of TA (CLS-TA, triamcinolone acetonide injectable suspension)
  Arms: 4 mg CLS-TA + IVT aflibercept
Drug: Sham — suprachoroidal sham procedure
  Other Names: suprachoroidal sham
  Arms: sham + IVT aflibercept
Drug: IVT aflibercept — 2 mg intravitreal injection of aflibercept
  Other Names: Eylea

SUMMARY:
A phase 2, multicenter, randomized, active-controlled, masked, parallel arm study designed to evaluate the safety and efficacy of a single suprachoroidal injection of CLS-TA, triamcinolone acetonide injectable suspension, given along with an intravitreal (IVT) injection of aflibercept compared to IVT aflibercept alone in subjects with retinal vein occlusion (RVO).

DETAILED DESCRIPTION:
A randomized, masked, controlled trial of safety and efficacy of suprachoroidal CLS-TA in combination with intravitreal aflibercept in subjects with macular edema following retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of macular edema following RVO
* History of ME ≤ 12 months
* 20-70 letters inclusive BCVA using ETDRS

Exclusion Criteria:

* has had an IVT injection of anti-VEGF for RVO in the study eye
* has had a corticosteroid injection in the past 3 months in the study eye
* any uncontrolled ophthalmic condition in the study eye other than RVO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical, Inc.
Locations (14):
- United States (14):
  - Phoenix, Arizona
  - Beverly Hills, California
  - San Diego, California
  - Boynton Beach, Florida
  - Atlanta, Georgia
  - Baltimore, Maryland
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Rapid City, South Dakota
  - Abilene, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - The Woodlands, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Suprachoroidal CLS-TA + IVT Aflibercept: Single unilateral, suprachoroidal injection of 40 mg/mL (4 mg in 100 µL) of CLS-TA following a 2 mg intravitreal injection of aflibercept
  suprachoroidal CLS-TA: suprachoroidal injection of CLS-TA
  IVT aflibercept: 2 mg intravitreal injection of aflibercept
- Suprachoroidal Sham + IVT Aflibercept: Single unilateral, suprachoroidal sham procedure following a 2 mg intravitreal injection of aflibercept
  suprachoroidal sham: suprachoroidal sham procedure
  IVT aflibercept: 2 mg intravitreal injection of aflibercept
Period: Overall Study
Arm/Group | Suprachoroidal CLS-TA + IVT Aflibercept | Suprachoroidal Sham + IVT Aflibercept
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat set included all randomly assigned subjects who were treated and had at least one post-Baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Suprachoroidal CLS-TA + IVT Aflibercept | Suprachoroidal Sham + IVT Aflibercept | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 18 | 13 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.9 (12.02) | 65.8 (14.64) | 66.3 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Times a Subject Qualifies to be Administered IVT Aflibercept in Each Arm
Time Frame: 3 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Suprachoroidal CLS-TA + IVT Aflibercept | Suprachoroidal Sham + IVT Aflibercept
Number analyzed (Participants) | 23 | 23
Participants
  0 | 18 | 7
  1 | 3 | 12
  2 | 0 | 1
  3 | 2 | 3

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Suprachoroidal CLS-TA + IVT Aflibercept | Suprachoroidal Sham + IVT Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 12/23 | 10/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suprachoroidal CLS-TA + IVT Aflibercept (N=23) | Suprachoroidal Sham + IVT Aflibercept (N=23)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Cataract (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 1 (1) — #Study eye
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 0 (0) — #Study eye
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Corneal oedema (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Eye pain (Eye disorders) | 8 (9) | 1 (1) — #Study eye
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Ocular discomfort (Eye disorders) | 0 (0) | 2 (2) — #Study eye
Ocular hypertension (Eye disorders) | 2 (2) | 0 (0) — #Study eye
Optic disc vascular disorder (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Retinal exudates (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Retinal haemorrhage (Eye disorders) | 1 (2) | 0 (0) — #Study eye
Retinopathy (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Vision blurred (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Vision blurred (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2) — #Study eye
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 0 (0) — #Study eye
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of Clearside.